CLINICAL TRIAL: NCT02795260
Title: Phase III Clinical Study of Recombinant Mycobacterium Tuberculosis Allergen ESAT6-CFP10 on Healthy People Aged 18-65,Adopting Randomized Blinded and Parallel Controlled Method
Brief Title: Clinical Study of Recombinant Mycobacterium Tuberculosis Allergen ESAT6-CFP10 on Healthy People Aged 18-65(III-healthy)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Anhui Zhifei Longcom Biologic Pharmacy Co., Ltd. (Industry)
Collaborators: Air Force Military Medical University, China (Other); Proswell Medical Corporation (Industry); Jiangsu Province Centers for Disease Control and Prevention (Network); Jurong Centers for Disease Control and Prevention (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: EC-III-healthy
Record Dates: First submitted 2016-03-14; First posted 2016-06-10 (Estimated); Last update posted 2020-10-01 (Actual); Status verified 2017-01

CONDITIONS: Tuberculosis
Keywords: ESAT6; CFP10; skin test; diagnostic test
MeSH Terms: conditions — Tuberculosis | interventions — BCG Vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ESAT6-CFP10 in the right arm (Experimental): Each volunteer is intradermally injected two agents in different arms 12 weeks after Bacillus Calmette - Guerin (BCG) or placebo of BCG immunization :ESAT6-CFP10 in the right arm and TB-PPD in the left arm concomitantly,according to a randomisation scheme.
  Interventions: Biological: Bacillus Calmette - Guerin; Biological: placebo of Bacillus Calmette - Guerin
- ESAT6-CFP10 in the left arm (Experimental): Each volunteer is intradermally injected two agents in different arms 12 weeks after Bacillus Calmette - Guerin (BCG) or placebo of Bacillus Calmette - Guerin immunization :ESAT6-CFP10 in the left arm and TB-PPD in the right arm concomitantly,according to a randomisation scheme.
  Interventions: Biological: Bacillus Calmette - Guerin; Biological: placebo of Bacillus Calmette - Guerin

INTERVENTIONS:
Biological: Bacillus Calmette - Guerin — The participants are injection intradermally with 0.1ml ESAT6-CFP10(EC) in the right OR left arm and TB-PPD in the other arm(right OR left) after 12 weeks immunization of BCG .
  Other Names: BCG
Biological: placebo of Bacillus Calmette - Guerin — The participants are injection intradermally with 0.1ml ESAT6-CFP10(EC) in the right OR left arm and TB-PPD in the other arm(right OR left) after 12 weeks immunization of placebo of BCG .
  Other Names: placebo of BCG

SUMMARY:
The investigators recruit about 1800 cases participants who has signed ICF,then do some physical examinations for these people, including ecg, X-ray, HIV,blood pressure, specific gamma-interferon detection ,collection of medical history and the like .These subjects who meet the standard are considered as study population I. Population I are injected intradermally with ESAT6-CFP10 and Tuberculin purified protein derivative(TB-PPD) at different arm of the same subject and get at least 360 participants whose three kinds of detection result are all negative and are considered as study population II.Then,they are immune to the Bacillus Calmette -Guerin(BCG) vaccine or the placebo of the BCG.Do specific gamma-interferon detection before the skin test,then inject intradermally with ESAT6-CFP10 and TB-PPD at different arm of the same subject 12 weeks after immunity.

DETAILED DESCRIPTION:
The investigators recruit about 1800 cases participants who has signed ICF,then do some physical examinations for these people, including ecg, X-ray, HIV,blood pressure, specific gamma-interferon detection(γ-IFN) ,collection of medical history and the like .These subjects who meet the standard are considered as study population I. Population I are injected intradermally with ESAT6-CFP10 and Tuberculin purified protein derivative(TB-PPD) at different arm of the same subject and get at least 360 participants whose three kinds of detection result are all negative(specific gamma-interferon detection ,TB-PPD and ESAT6-CFP10 ) and are considered as study population II.Then,they are immune to the Bacillus Calmette -Guerin(BCG) vaccine or the placebo of the BCG(BCG and the palcebo ratio of 2:1 ),they are incorporated into the Population III. Do specific gamma-interferon detection before the skin test,then inject intradermally with ESAT6-CFP10 and TB-PPD at different arm of the same subject 12 weeks after immunity. Evaluate the specificity of the ESAT6-CFP10 allergen by negative coincidence rate for BCG vaccinated crowd ,and the safety of ESAT6-CFP10 in all participant,and the correlation between ESAT6-CFP10 ,TB-PPD and γ-IFN.

ELIGIBILITY:
Inclusion Criteria of the screening crowd

1. 18-65 years old;
2. consent and signed informed consent form;
3. comply with follow-up;
4. No history of tuberculosis;
5. Physical condition:no obvious heart,liver,kidney, digestive tract,nervous system,mental disorder from signed informed consent to the injection;
6. Normal axillary temperature (quiet condition blow 37.0℃)
7. No abnormal chest by X-ray check;

Exclusion Criteria of the screening crowd

1. Has the following serious disease, such as advanced cancer, diabetes, chronic obstructive pulmonary disease (copd) in acute episodes, acute/ progressive liver disease or kidney disease, congestive heart failure, etc;
2. Epilepsy and psychiatric patients
3. Has known or suspected (or risk possible) immune damaged or abnormal functional , accept glucocorticoid and immunosuppressants or immunopotentiator treatment, outside the gastrointestinal tract protein or blood products or plasma extraction in 3 months；
4. Has acute febrile diseases and infectious diseases;
5. taking part in any other new drug clinical trials or participated in any other new drug clinical trials within 3 months before this trials;
6. a clear history of drug allergy ；
7. In pregnancy or lactation；
8. There is a clear history of high blood pressure and systolic blood pressure ≥180mmHg , and/or diastolic blood pressure of ≥ 100mmHg after drug control ；
9. Researchers consider that any conditions may affect the trial evaluation.

Inclusion Criteria of three negative crowd

1. conforming to the inclusion criteria of the screening crowd ;
2. the result of four detection methods are all the negative: ESAT6-CFP10 、 TB - PPD and specific gamma - IFN and HIV;

Exclusion Criteria of three negative crowd

1. conforming to the exclusion criteria of the screening crowd ;
2. With BCG vaccination taboo .

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1802 (Actual)
Dates: Start 2016-05; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Number of study population III Negative for Reaction at 24 hours After intradermal injection with EC or TB-PPD | At 24 hours after Intradermal injection with EC or TB-PPD
Number of study population III Negative for Reaction at 48 hours After intradermal injection with EC or TB-PPD | At 48 hours after Intradermal injection with EC or TB-PPD

SECONDARY OUTCOMES:
the number of participants with Adverse Events after Intradermal injection | within 48 hours after after Intradermal injection

CONTACTS AND LOCATIONS:
Overall Officials: Wei Lu, Master, Principal Investigator — Jiangsu Province Centers for Disease Control and Prevention

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ravn P, Munk ME, Andersen AB, Lundgren B, Lundgren JD, Nielsen LN, Kok-Jensen A, Andersen P, Weldingh K. Prospective evaluation of a whole-blood test using Mycobacterium tuberculosis-specific antigens ESAT-6 and CFP-10 for diagnosis of active tuberculosis. Clin Diagn Lab Immunol. 2005 Apr;12(4):491-6. doi: 10.1128/CDLI.12.4.491-496.2005. PMID 15817755
- [Background] Brusasca PN, Colangeli R, Lyashchenko KP, Zhao X, Vogelstein M, Spencer JS, McMurray DN, Gennaro ML. Immunological characterization of antigens encoded by the RD1 region of the Mycobacterium tuberculosis genome. Scand J Immunol. 2001 Nov;54(5):448-52. doi: 10.1046/j.1365-3083.2001.00975.x. PMID 11696195
- [Background] Weldingh K, Andersen P. ESAT-6/CFP10 skin test predicts disease in M. tuberculosis-infected guinea pigs. PLoS One. 2008 Apr 23;3(4):e1978. doi: 10.1371/journal.pone.0001978. PMID 18431468
- [Background] Aagaard C, Govaerts M, Meikle V, Vallecillo AJ, Gutierrez-Pabello JA, Suarez-Guemes F, McNair J, Cataldi A, Espitia C, Andersen P, Pollock JM. Optimizing antigen cocktails for detection of Mycobacterium bovis in herds with different prevalences of bovine tuberculosis: ESAT6-CFP10 mixture shows optimal sensitivity and specificity. J Clin Microbiol. 2006 Dec;44(12):4326-35. doi: 10.1128/JCM.01184-06. Epub 2006 Sep 27. PMID 17005738
- See also: CENTER FOR DRUG EVALUATION,NMPA — http://www.cde.org.cn/